CLINICAL TRIAL: NCT04178668
Title: Molecular and Organizational Changes in the Human Oral Mucosa During Aging
Acronym: MMOBUCC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in recruitment
Sponsor: University Hospital, Toulouse (Other)
Collaborators: University Paul Sabatier of Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC31/19/0423
Record Dates: First submitted 2019-11-13; First posted 2019-11-26 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Oral Health
Keywords: molecular mobility; collagen denaturation; oral mucosa; saliva; ageing
MeSH Terms: interventions — Endomet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 20-40 years old (Experimental): 33 patients between 20 and 40 years old
  Interventions: Other: Oral mucosa and saliva samples
- 70-90 years old (Experimental): 33 patients between 70 and 90 years old
  Interventions: Other: Oral mucosa and saliva samples

INTERVENTIONS:
Other: Oral mucosa and saliva samples — one oral mucosa sample and one saliva sample

SUMMARY:
The objective of this interventional with mucosa et saliva samples, monocentric, transversal and pilot study is to extract vibrational, thermal and dielectric markers obtained by Differential Scanning Calorimetry, Thermo-Stimulated Currents and Fourier Transform Infrared spectroscopy on oral mucosa and saliva samples collected from 66 patients divided in two groups (20-40 and 70-90 years old).

DETAILED DESCRIPTION:
Edentulism is prevalent in elderly people and the current care is the use of removable denture based on edentulous jaw regions. Nevertheless, the close and extended contact of denture base with mucosa and the transmission of chewing movement trough the complete denture leads to a weakening of supporting tissues in the medium to long term. This embrittlement may be accompanied by pain, compromising the proper integration of complete denture. In geriatrics, the peculiar weakness of bearing surfaces, connected to physio-pathological conditions as well as the decrease of adaptability and resistance further complicate the biomechanical integration of this kind of prosthesis. It has been shown that chronical ageing induces a decrease of resiliency and hydration of oral mucosa, associated with a decrease of epithelium thickness; nevertheless few studies have been performed at the molecular and supramolecular level to characterize this mucosa. Techniques of material characterization (Fourier transform Infrared spectroscopy, Differential scanning calorimetry (DSC), Thermostimulated currents (TSC), have shown their ability to follow hydric, molecular and structural modification of dermis upon ageing. In accordance with this study, the distribution of thermal, vibrational and dielectric markers of oral mucosa will be extracted in two age groups. The principal hypothesis of the research is the possibility to identify specific markers and to follow molecular and organizational changes induced by ageing (intrinsic ageing or extrinsic ageing due to prostheses wearing). The characterization of saliva by Fourier transform infrared spectroscopy (FTIR) shows promise in quantifying the biochemical components of this biofluid. Some vibrational saliva biomarkers have high diagnostic potential (physiological stress, diabetes, salivary lithiasis, carcinomas, periodontitis).This study is a first step to redefine the specification for the most appropriate biomaterial in removable prostheses.

ELIGIBILITY:
Inclusion Criteria:

* Patient requiring a classic dental surgery (extraction, implantology...) at the Toulouse University Hospital,
* Between the ages of 20 and 40 or between 70 and 90 years

Exclusion Criteria:

* Patient with gastrotomy probes or chemotherapy, palliative care (or with a life expectancy of less than 30 days),
* Patient with surgical contraindication: allergy to local anesthetics, major hemorrhagic risk: patient on unbalanced Anti Vitamin K, patient on new anticoagulants not relayed or not discontinued,
* Patient at high risk of infectious endocarditis
* Patient under safeguard of justice.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2021-10-27 (Actual)

PRIMARY OUTCOMES:
Vibrational marker of the oral mucosa: collagen 1 fraction indicator | Day 0
  collagen 1 fraction indicator measured by Fourier-transform infrared spectroscopy. It corresponds to the ratio of the band area 1338 cm-1/1750-1000 cm-1
Vibrational marker of the oral mucosa : collagen 2 fraction indicator | Day 0
  collagen 2 fraction indicator measured by Fourier-transform infrared spectroscopy. It corresponds to the ratio of the band area 1202 cm-1/1750-1000 cm-1
Thermal marker of the oral mucosa : percentage of open water | Day 0
  percentage of open water
Thermal marker of the oral mucosa: percentage of water related | Day 0
  percentage of water related
Thermal marker of the oral mucosa : percentage of total water | Day 0
  percentage of total water
Thermal marker of the oral mucosa : maximum denaturation temperature | Day 0
  maximum denaturation temperature
Thermal marker of the oral mucosa : collagen denaturation enthalpy | Day 0
  collagen denaturation enthalpy (in J/g) determined by differential calorimetric analysis
Dielectric marker of the oral mucosa : temperature of mode 1 in the hydrated state | Day 0
  temperature of mode 1 in the hydrated state

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Hélène LACOSTE-FERRE, MD, Principal Investigator — University Hospital of Toulouse
Locations (1):
- University hospital of Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lacoste-Ferre MH, Ober C, Samouillan V. Viscoelastic behavior of oral mucosa. A rheological study using small-amplitude oscillatory shear tests. J Mech Behav Biomed Mater. 2023 Jul;143:105898. doi: 10.1016/j.jmbbm.2023.105898. Epub 2023 May 5. PMID 37156074